CLINICAL TRIAL: NCT01404689
Title: Midazolam With Meperidine and Dexmedetomidine vs Midazolam With Meperidine for Sedation During ERCP
Brief Title: Study to Determine if the Midazolam-Meperidine-Dexmedetomidine is Superior to the Midazolam-Meperidine for Sedation During ERCP
Acronym: DEMMER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Hana Pharm Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Sang Hyub Lee, Assistant Professor of Internal Medicine, Seoul National University College of Medicine and Seoul National University Bundang Hospital, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SNUBH-129-012
Record Dates: First submitted 2011-07-24; First posted 2011-07-28 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Undergoing ERCP for Diagnostic or Therapeutic Purposes
Keywords: dexmedetomidine; midazolam; ERCP; cholangiopancreatography; sedation; propofol
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Midazolam-Meperidine-Dexmedetomidine (Experimental): midazolam 0.06mg/kg IV bolus, meperidine 50mg IV bolus and dexmedetomidine 1μg/Kg•hr infusion (30% reduction of midazolam dose and 25mg of meperidine for patients 65 years of age or older)
  Interventions: Drug: Dexmedetomidine
- Midazolam-Meperidine (Sham Comparator): midazolam 0.06mg/kg IV bolus, meperidine 50mg IV bolus and placebo(saline) infusion(30% reduction of midazolam dose and 25mg of meperidine for patients 65 years of age or older)
  Interventions: Other: normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — dexmedetomidine 1μg/Kg•hr IV continuous infusion, initiated 15 min before the procedure (ERCP) till complete procedure
  Other Names: Precedex® 100μg/1ml vial: DMDTIA
  Arms: Midazolam-Meperidine-Dexmedetomidine
Other: normal saline — 0.9% NaCl 1μg/Kg•hr IV continuous infusion, initiated 15 min before the procedure (ERCP) till complete procedure
  Other Names: NaCl 0.9% 20ml plastic ample: NSIP
  Arms: Midazolam-Meperidine

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) takes a longer time and is more complex to perform than the other parallel procedures, causing discomfort to patients. It is commonly performed under sedation endoscopy. Until recently, the combination administration of midazolam and opioid has been widely used as standard therapy due to its superior sedation effect compared to the other sedation agents. Midazolam, however, has problems, such as an insufficient sedation effect and an intermittent paradoxical response.

Unlike midazolam, propofol has no antagonist and may cause problems such as respiratory depression, and has a narrow therapeutic range for the sedation effect, consequently requiring supervision by experienced experts, although it has a better sedation effect than midazolam. Due to these disadvantages, propofol is clinically less useful than midazolam.

Meanwhile, dexmedetomidine, a selective α2 adrenergic agonist, is known to maintain the proper level of sedation and has a weak influence on respiratory depression. Recent studies have shown positive results with dexmedetomidine in relation with the sedation effect for surgery patients under local anesthesia or in intensive care units.

As such, extensive studies are being conducted on the use of dexmedetomidine in endoscopic procedures due to the increased attention to dexmedetomidine. This notwithstanding, the clinical usefulness of dexmedetomidine is still debatable. In particular, studies on the use of dexmedetomidine for ERCP are very rare.

Given the recent idea that dexmedetomidine may exert a synergistic effect in combination with midazolam, these authors endeavored to prospectively compare and analyze the sedation effect and adverse events, including respiratory depression, of the combination therapy of midazolam and meperidine, both of which have been widely used in patients undergoing ERCP, and of the combination therapy of midazolam, meperidine, and dexmedetomidine.

The small-scale comparative study on the combination administration of propofol and fentanyl, which has a high risk of causing complications, and on the single administration of dexmedetomidine is the only study on the sedation effect of dexmedetomidine in the ERCP procedure that has yet been conducted; there has been no study that investigated the effect of the combination administration of dexmedetomidine and other drugs in the ERCP procedure. This study is thus expected to contribute to the development of guidelines on sedation in the ERCP procedure.

DETAILED DESCRIPTION:
Compared with upper gastrointestinal endoscopy, endoscopic retrograde cholangiopancreatography (ERCP) takes a longer time to perform and causes more discomfort to patients. In ERCP, benzodiazepine alone or in combination with opioid is commonly used for pain control and sedation.

Of the various benzodiazepine drugs, midazolam, which is water-soluble, has been shown to act faster and to be better in terms of anterograde amnesia and its sedation effect than other drugs. As midazolam has a suitable antagonist (flumazenil), prompt measures can be taken in case of such situations as hypopnea.

As midazolam was reported to increase the sedation effect and the level of satisfaction of patients when used in combination with opioid (meperidine), a combination of midazolam and meperidine has been the most widely used regimen so far. The American Society for Gastrointestinal Endoscopy recommends a combination of midazolam and meperidine as a standard regimen for inducing sedation in upper and lower gastrointestinal endoscopy.

Several studies reported, however, that midazolam alone or the combination of midazolam and meperidine was insufficient for inducing the sedation effect (47-80%). Besides, midazolam has the disadvantage of producing a paradoxical response at times, which makes the performance of the procedure impossible.

In many studies, propofol, which is preferred as an alternative to midazolam, was recently found to be superior to midazolam in terms of its sedation effect, as it does not cause adverse events.

Because propofol intermittently causes serious respiratory failure and has no antagonist, however, clinicians feel burdened with the use of propofol, due to which it is not widely used. Moreover, anesthesia specialists as well as experienced assistant staff who had received relevant education and training should be available, and all tools needed to promptly handle cardiopulmonary complications should be on hand, which lowers the usefulness of propofol in clinical practice.

The sedation effect of dexmedetomidine, however, a selective α2 adrenergic receptor, is proportional to its dose, so it allows continuous injection and makes it possible to reduce the opioid dose needed for sedation when it is used for sedation. Dexmedetomidine was reported to maintain a proper level of sedation, and to influence less the respiratory rate, oxygen saturation, and respiratory tract response. Due to these advantages, several recent studies reported that dexmedetomidine can be effective for sedation during upper and lower gastrointestinal procedures.

A combination of dexmedetomidine and midazolam was investigated in recent trials with animals and in clinical trials, and its synergic effect was shown in several studies.

In an animal trial using rats, Boehm et al. reported that midazolam increased the dose-related analgesic effect of dexmedetomidine when it was used in combination with dexmedetomidine. Bol et al. reported that combined administration of dexmedetomidine and midazolam increased the sedation effect while reducing adverse cardiovascular events more significantly than with a single administration.

In addition, in a study on rats, Salonen et al. demonstrated the synergic effect of the combination of the two drugs and that flumazenil antagonized the combination of the two drugs in a dose-dependent manner.

In one of the representative clinical trials, Bergese et al. compared a combination of dexmedetomidine and midazolam with a midazolam-alone regimen in 55 patients who underwent awake fibrotic intubation (AFOI).

Although there was no hemodynamic difference between the two groups, the combination regimen had a better sedation effect, resulted in a higher level of satisfaction among the patients, and led to fewer adverse events than did the single regimen.

Besides, in a study on patients who underwent cardiovascular surgery, Dasta et al. reported that the use of dexmedetomidine in combination with a standard sedation regimen decreased mortality and reduced the period of mechanical ventilation and the cost. Heard et al. reported that combined administration of midazolam and dexmedetomidine had a sufficient sedation effect on patients who had undergone MRI without adverse events. In the study by Heard et al.,however, in which the subjects were children, propofol was used as the control drug instead of midazolam.

So far, no studies have reported the effect of combination administration of dexmedetomidine and midazolam in gastrointestinal endoscopy, including in ERCP. Given the synergic effect of the two drugs and the usefulness of dexmedetomidine in endoscopy, such studies are urgently needed.

Though the study by Muller et al. was not on the effect of the combined administration, it is the only study that investigated the sedation effect of dexmedetomidine in ERCP.

In the study by Muller et al. on 26 patients who had undergone ERCP (12 of whom received dexmedetomidine and 14, propofol), they reported that the effect of sedation and pain control was weaker in the dexmedetomidine group than in the propofol group (RR: 2.71/9.42 and NNT: 1.85/1.42, respectively), and that the hemodynamic instability was high in the dexmedetomidine group based on the subjects' mean blood pressure and the heart rate.

The study by Muller et al. had limitations, however, in that the dose of dexmedetomidine was lower than that in other studies and the scale of the study was small. Moreover, although the mean blood pressure and the heart rate were lower in the dexmedetomidine group than in the propofol group, no clinically significant decrease in the blood pressure and the heart rate was observed.

Moreover, propofol, which was used in the control group, may impose a heavy burden in relation to its depressing respiratory effect because of the absence of an antagonist (flumazenil), unlike with midazolam, as described previously, which acts faster and requires experienced assistant staff; and because the usefulness and frequency of use of propofol in clinical practice is low. In addition, as the study by Muller et al. was about single dexmedetomidine administration, the comparison of the combined administration of dexmedetomidine and midazolam with the single administration of propofol to produce the sedation effect could result in different outcomes.

As such, it is believed that the sedation effect and adverse events from the combined administration of dexmedetomidine and midazolam and from single administration of midazolam in patients who had undergone ERCP should be studied.

As described previously, midazolam is considered suitable as a control drug as it is more useful than propofol in clinical practice. Moreover, since the combination of dexmedetomidine and midazolam has a synergic effect on sedation, the combination is believed to be more meaningful than single dexmedetomidine administration.

In addition, the cardiovascular and respiratory safety of single dexmedetomidine administration and the combined administration of dexmedetomidine and midazolam, as reported in several previous studies, was shown as satisfactory in this study.

Whether or not this synergic effect and safety will be seen as well in gastrointestinal endoscopy, particularly in ERCP, will be further investigated; and as there is no study yet that has investigated the combined administration of dexmedetomidine and midazolam in patients undergoing ERCP, this study can be considered meaningful.

ELIGIBILITY:
Inclusion Criteria:

* Those who are admitted for diagnostic and therapeutic ERCPs
* aged 20 to 80 years
* American Society of Anesthesiologists (ASA) classification I to III

Exclusion Criteria:

* ASA physical status IV and V
* allergic to any components of sedation and opioid drugs
* patients with chronic illicit drug use

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Level of sedation | During entire procedure(ERCP) time; an expected average of the procedure time is 20 minutes
  The sedation level recorded by the RSS and the requirement of the additional sedative (midazolam) or the analgesic (meperidine), and the proportion (%) of cases where adequate sedation was maintained during entire procedure time.

SECONDARY OUTCOMES:
Complication rate | From start point of the procedure(ERCP) to 60 minutes after the procedure
  * Change in respiration and hemodynamics
    * Mean blood pressure
    * Heart rate
    * Respiratory rate
    * Oxygen saturation
  * Adverse effects
  * The procedure and discharge time
  * Pain and patient satisfaction
  * Bispectral index scores

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hyub Lee, M.D. Ph.D, Study Director — Assistant Professor of Internal Medicine, Seoul National University College of Medicine and Seoul National University Bundang Hospital; Ban Seok Lee, M.D., Principal Investigator — Fellowship doctor, Division of Gastroenterology, Department of Internal Medicine, Seoul National University Bundang Hospital
Locations (1):
- Division of Gastroenterology, Department of Internal Medicine, Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Background] Standards of Practice Committee of the American Society for Gastrointestinal Endoscopy; Lichtenstein DR, Jagannath S, Baron TH, Anderson MA, Banerjee S, Dominitz JA, Fanelli RD, Gan SI, Harrison ME, Ikenberry SO, Shen B, Stewart L, Khan K, Vargo JJ. Sedation and anesthesia in GI endoscopy. Gastrointest Endosc. 2008 Nov;68(5):815-26. doi: 10.1016/j.gie.2008.09.029. No abstract available. PMID 18984096
- [Background] Yuksel O, Parlak E, Koklu S, Ertugrul I, Tunc B, Sahin B. Conscious sedation during endoscopic retrograde cholangiopancreatography: midazolam or midazolam plus meperidine? Eur J Gastroenterol Hepatol. 2007 Nov;19(11):1002-6. doi: 10.1097/MEG.0b013e3282cf5167. PMID 18049171
- [Background] Reimann FM, Samson U, Derad I, Fuchs M, Schiefer B, Stange EF. Synergistic sedation with low-dose midazolam and propofol for colonoscopies. Endoscopy. 2000 Mar;32(3):239-44. doi: 10.1055/s-2000-134. PMID 10718390
- [Background] Honan VJ. Paradoxical reaction to midazolam and control with flumazenil. Gastrointest Endosc. 1994 Jan-Feb;40(1):86-8. doi: 10.1016/s0016-5107(94)70020-6. No abstract available. PMID 8163147
- [Background] Chen WX, Lin HJ, Zhang WF, Gu Q, Zhong XQ, Yu CH, Li YM, Gu ZY. Sedation and safety of propofol for therapeutic endoscopic retrograde cholangiopancreatography. Hepatobiliary Pancreat Dis Int. 2005 Aug;4(3):437-40. PMID 16109532
- [Background] Kongkam P, Rerknimitr R, Punyathavorn S, Sitthi-Amorn C, Ponauthai Y, Prempracha N, Kullavanijaya P. Propofol infusion versus intermittent meperidine and midazolam injection for conscious sedation in ERCP. J Gastrointestin Liver Dis. 2008 Sep;17(3):291-7. PMID 18836622
- [Background] Ladas SD, Aabakken L, Rey JF, Nowak A, Zakaria S, Adamonis K, Amrani N, Bergman JJ, Boix Valverde J, Boyacioglu S, Cremers I, Crowe J, Deprez P, Dite P, Eisen M, Eliakim R, Fedorov ED, Galkova Z, Gyokeres T, Heuss LT, Husic-Selimovic A, Khediri F, Kuznetsov K, Marek T, Munoz-Navas M, Napoleon B, Niemela S, Pascu O, Perisic N, Pulanic R, Ricci E, Schreiber F, Svendsen LB, Sweidan W, Sylvan A, Teague R, Tryfonos M, Urbain D, Weber J, Zavoral M; European Society of Gastrointestinal Endoscopy Survey of National Endoscopy Society Members. Use of sedation for routine diagnostic upper gastrointestinal endoscopy: a European Society of Gastrointestinal Endoscopy Survey of National Endoscopy Society Members. Digestion. 2006;74(2):69-77. doi: 10.1159/000097466. Epub 2006 Nov 27. PMID 17135728
- [Background] Cohen LB, Delegge MH, Aisenberg J, Brill JV, Inadomi JM, Kochman ML, Piorkowski JD Jr; AGA Institute. AGA Institute review of endoscopic sedation. Gastroenterology. 2007 Aug;133(2):675-701. doi: 10.1053/j.gastro.2007.06.002. No abstract available. PMID 17681185
- [Background] Kamibayashi T, Maze M. Clinical uses of alpha2 -adrenergic agonists. Anesthesiology. 2000 Nov;93(5):1345-9. doi: 10.1097/00000542-200011000-00030. No abstract available. PMID 11046225
- [Background] Kunisawa T, Hanada S, Kurosawa A, Suzuki A, Takahata O, Iwasaki H. Dexmedetomidine was safely used for sedation during spinal anesthesia in a very elderly patient. J Anesth. 2010 Dec;24(6):938-41. doi: 10.1007/s00540-010-1025-z. Epub 2010 Oct 7. PMID 21110048
- [Background] Dere K, Sucullu I, Budak ET, Yeyen S, Filiz AI, Ozkan S, Dagli G. A comparison of dexmedetomidine versus midazolam for sedation, pain and hemodynamic control, during colonoscopy under conscious sedation. Eur J Anaesthesiol. 2010 Jul;27(7):648-52. doi: 10.1097/EJA.0b013e3283347bfe. PMID 20531094
- [Background] Boehm CA, Carney EL, Tallarida RJ, Wilson RP. Midazolam enhances the analgesic properties of dexmedetomidine in the rat. Vet Anaesth Analg. 2010 Nov;37(6):550-6. doi: 10.1111/j.1467-2995.2010.00565.x. PMID 21040379
- [Background] Bol CJ, Vogelaar JP, Tang JP, Mandema JW. Quantification of pharmacodynamic interactions between dexmedetomidine and midazolam in the rat. J Pharmacol Exp Ther. 2000 Jul;294(1):347-55. PMID 10871332
- [Background] Salonen M, Onaivi ES, Maze M. Dexmedetomidine synergism with midazolam in the elevated plus-maze test in rats. Psychopharmacology (Berl). 1992;108(1-2):229-34. doi: 10.1007/BF02245313. PMID 1357706
- [Background] Bergese SD, Patrick Bender S, McSweeney TD, Fernandez S, Dzwonczyk R, Sage K. A comparative study of dexmedetomidine with midazolam and midazolam alone for sedation during elective awake fiberoptic intubation. J Clin Anesth. 2010 Feb;22(1):35-40. doi: 10.1016/j.jclinane.2009.02.016. PMID 20206849
- [Background] Dasta JF, Jacobi J, Sesti AM, McLaughlin TP. Addition of dexmedetomidine to standard sedation regimens after cardiac surgery: an outcomes analysis. Pharmacotherapy. 2006 Jun;26(6):798-805. doi: 10.1592/phco.26.6.798. PMID 16716133
- [Background] Heard C, Burrows F, Johnson K, Joshi P, Houck J, Lerman J. A comparison of dexmedetomidine-midazolam with propofol for maintenance of anesthesia in children undergoing magnetic resonance imaging. Anesth Analg. 2008 Dec;107(6):1832-9. doi: 10.1213/ane.0b013e31818874ee. PMID 19020127
- [Background] Muller S, Borowics SM, Fortis EA, Stefani LC, Soares G, Maguilnik I, Breyer HP, Hidalgo MP, Caumo W. Clinical efficacy of dexmedetomidine alone is less than propofol for conscious sedation during ERCP. Gastrointest Endosc. 2008 Apr;67(4):651-9. doi: 10.1016/j.gie.2007.09.041. Epub 2008 Mar 4. PMID 18291396
- [Derived] Lee BS, Ryu J, Lee SH, Lee MG, Jang SE, Hwang JH, Ryu JK, Do SH, Kim YT. Midazolam with meperidine and dexmedetomidine vs. midazolam with meperidine for sedation during ERCP: prospective, randomized, double-blinded trial. Endoscopy. 2014 Apr;46(4):291-8. doi: 10.1055/s-0033-1358909. Epub 2014 Mar 26. PMID 24671858
- See also: Web site of Seoul National University Bundang Hospital — http://www.snubh.org/
- See also: Web site of Seoul National University College of Medicine — http://medicine.snu.ac.kr/
- See also: Web site of Korea Food and Drug Administration — http://www.kfda.go.kr/